CLINICAL TRIAL: NCT02272504
Title: A Randomized Controlled Trial to Determine the Role of Biomarkers in Surveillance for Hepatocellular Carcinoma (HCC)
Brief Title: A Protocol of the Canadian Prospective Study for Hepatocellular Carcinoma Surveillance Using Biomarkers
Status: Completed | Type: Observational
Sponsor: Wako Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: WLS 13-6926
Record Dates: First submitted 2014-10-20; First posted 2014-10-23 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Cirrhosis; Chronic Liver Diseases
Keywords: HCC; AFP; AFP-L3; DCP; Surveillance; biomarkers
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen Serum samples will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Standard of care arm: Chronic liver disease patients who are under going standard of care surveillance for the development of HCC as defined by AASLD guidelines.
- Biomarker Arm: Chronic liver disease patients who are under going standard of care surveillance for the development of HCC as defined by AASLD guidelines plus the addition of biomarker assays (AFP, AFP-L3 and DCP) every 6 months.

SUMMARY:
The objective of this study is to evaluate the clinical effectiveness of biomarkers, alpha-fetoprotein (AFP), Lens culinaris agglutinin-reactive fraction of AFP (AFP-L3), and des-gamma-carboxy prothrombin (DCP), for surveillance program patients whose hepatocellular carcinoma (HCC) development may be potentially missed by ultrasound (US). This study expects to demonstrate that addition of biomarkers will increase the detection rate by at least 10%.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial (RCT) comparing surveillance for hepatocellular carcinoma with ultrasound alone versus ultrasound and standard biomarkers. The study will be conducted initially at UHN (TGH and TWH). One arm will undergo surveillance for hepatocellular carcinoma using ultrasound (US) alone and the other will undergo HCC surveillance with US plus biomarkers (BM). The biomarkers to be used will be AFP, AFP-L3 and DCP). Subjects will undergo surveillance at 6 monthly intervals for a minimum of 2 years and up to 4 years. The endpoints will be the comparative effectiveness, defined as sensitivity and specificity of detection of HCC. The comparisons of sensitivity, specificity, and other parameters with respect to tumor characteristics will be made among US alone, biomarkers alone, and combined use of US and biomarkers. The target population is individuals who have liver cirrhosis and no HCC detectable at enrollment into the study. The factors contributing to the cause of the cirrhosis will be recorded but will not play a role into subject eligibility for the study

ELIGIBILITY:
Inclusion Criteria:

* Patient who is able and willing to comply with study procedures, and signed and dated informed consent is obtained.

  * Patients with a clinical suspicion of cirrhosis based on the investigator's evaluation with cirrhosis confirmed by one of the following: (see below for definition of cirrhosis). Etiology of cirrhosis will not be considered in determining inclusion in the study.
  * Patients aged 18 years and older.
  * Hep B Risk Score > 8 (table 1)

Table 1 Variable Risk Score Variable Risk Score Male 2 ALT <15 0 Female 0 ALT 15-44 1 Age 30-34 0 ALT > 45 2 Age 35-39 1 HBeAg+ve 0 Age 40-44 2 Anti-HBe-positive 2 Age 45-49 3 HBV DNA <300 copies/mL 0 Age 50-54 4 HBV DNA 300-9999 copies/mL 0 Age 55-59 5 HBV DNA 104 -99,000 copies/mL 3 Age 60-65 6 HBV DNA 105 - 999,999 copies/mL 5 HBV DNA > 106 copies/mL 4

Exclusion Criteria:

* • Patients who have confirmed HCC by CT/MRI when they enrolled. Patients who have previously had HCC but have been treated and have been recurrence free for 5 years are eligible.

  * Patients with the other cancer(s)
  * Pregnant Women
  * Patients who have known diagnosis of mental incapacitation that affects their ability to consent.
  * Patients who are likely to be transplanted within 1 year or MELD score greater than 20.
  * Patients with total or direct bilirubin > 3x upper limit of normal
  * Patients with uncontrollable ascites
  * Glomerular Filtration Rate less than 60.
  * Patients with ≥ Grade II of hepatic encephalopathy
  * Patients who are being treated with warfarin (DCP test values are affected by warfarin)
  * Patients who have any contraindication to any of the study procedures, products used or its constituents (e.g., renal failure or contrast allergy).
  * Patients who suffer from claustrophobia or who have other contraindications to MRI
  * Patients with cirrhosis who were successfully treated for hepatitis C more than 3 years prior. However, patients who are on study who are treated for their hepatitis C may continue in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at risk for the development of HCC as identified by the prior presence of chronic liver disease and cirrhosis.
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2014-08; Primary Completion 2020-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Biomarker assays exceeding threshold | Every 6 months until HCC is detected or up to 4 years
  Biomarker assay levels that exceed threshold will trigger diagnostic imaging for HCC. Ultrasound imaging indicating a suspicious nodule may also trigger diagnostic imaging.

SECONDARY OUTCOMES:
Surveillance until HCC development and detection | Up to 4 years
  When the total number of HCC cases as diagnosed by CT/MRI have been observed. Approximately 300 cases in total half (150) the cases from each group

CONTACTS AND LOCATIONS:
Overall Officials: Feld Jordan, MD, Principal Investigator — Toronto General Hospital
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Hirode G, Zangneh HF, Cerocchi O, Khalili K, El-Karim LA, Kandel C, Vecchio M, Winick J, Mori Y, Yamada H, Janssen HLA, Hansen BE, Sherman M, Feld JJ. Utility of Serum Biomarkers in Addition to Ultrasound for Early Detection of Hepatocellular Carcinoma in High-Risk Patients: A Randomized Controlled Trial. Gastroenterology. 2026 Jan 20:S0016-5085(25)05993-1. doi: 10.1053/j.gastro.2025.09.010. Online ahead of print. PMID 41556856